CLINICAL TRIAL: NCT04553627
Title: Allergan IIT-2019-10713 Feasibility of Producing the Appearance of a Gluteal Lift Post Cryolipolysis
Brief Title: Feasibility of Producing the Appearance of a Gluteal Lift Post Cryolipolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riverchase Dermatology (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allergan IIT-2019-10713
Record Dates: First submitted 2020-07-31; First posted 2020-09-17 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Subcutaneous Fat
Keywords: reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional cohort (Experimental): Zeltiq system is a thermoelectric device that applies controlled cooling ot skin. The CoolAdvantage applicators use gentle vacuum pressure to draw tissue into the cup shaped applicator. A gelpad is applied to skin to improve thermal coupling between participant and the applicator cooling surface.
  Interventions: Device: ZELTIQ thermoelectric device

INTERVENTIONS:
Device: ZELTIQ thermoelectric device — This is a feasibility study to determine if cryolipolysis in this area produces a desirable lifted appearance to the buttocks. Typically, a lifted more youthful appearance is obtained through surgical means. Study participants will be recruited from the population of patients who have suitable, treatable subcutaneous fat on the medial infragluteal folds and desire a lifted appearance. Subjects will receive treatments with a cooled cup cryolipolysis applicator from the CoolAdvantage family of applicators (cooled cup vacuum applicator). Treatments will be performed with a treatment temperature of - 11°C for up to 35 minutes. Subjects will complete all study-required follow-up visits, including an 8-week follow-up which may include a second treatment session, as well as a 12-week post final treatment follow-up visit

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of cryolipolysis of the medial infragluteal fold to create the appearance of a gluteal lift.

DETAILED DESCRIPTION:
In this study, the safety and the efficacy of ZELTIQ's technology will be evaluated for the non-invasive fat reduction of the medial infragluteal folds on a small group of subjects. This is a feasibility study to determine if cryolipolysis in this area produces a desirable lifted appearance to the buttocks. Typically, a lifted more youthful appearance is obtained through surgical means. Study participants will be recruited from the population of patients who have suitable, treatable subcutaneous fat on the medial infragluteal folds and desire a lifted appearance. Subjects will receive treatments with a cooled cup cryolipolysis applicator from the CoolAdvantage family of applicators (cooled cup vacuum applicator). Treatments will be performed with a treatment temperature of - 11°C for up to 35 minutes. Subjects will complete all study-required follow-up visits, including an 8-week follow-up which may include a second treatment session, as well as a 12-week post final treatment follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects > 22 years of age and < 50 years of age.
* Presence of suitable treatable subcutaneous fat on the medial infragluteal folds, which in the investigator's opinion may benefit from CoolSculpting to potentially create a lifted appearance to the buttocks.
* BMI under 30.
* No weight change exceeding 5% of body weight in the preceding month.
* Agreement to maintain their weight (i.e., within 5%) by not making any major changes in their diet or lifestyle during the course of the study.
* Subject has read and signed a written informed consent form

Exclusion Criteria:

* Subject has skin laxity in the area of intended treatment which in the opinion of the investigator, may result in an unacceptable aesthetic result.
* Subject has had a surgical procedure(s) in the area of intended treatment.
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.), in or around the area of intended treatment.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars, infection, in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Subject has a history of hernia in the areas to be treated.
* Pregnant or intending to become pregnant in the next 5 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female subjects > 22 years of age and < 50 years of age will be selected for this feasibility assessment
Enrollment: 10 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events [Safety and Tolerability] | 12 weeks
  The primary endpoint of the study is to evaluate the safety of subcutaneous fat reduction in the medial intragluteal folds using the ZELTIQ System as a non-invasive clinical treatment. Safety will be measured through the incidence of device and/or procedure-related adverse event.
Subjective clinical evaluation of subcutaneous fat treatment by Cryolipolysis [Efficacy] | 12 weeks
  The primary endpoint of the study is to evaluate the efficacy of subcutaneous fat reduction in the medial intragluteal folds using the ZELTIQ System as a non-invasive clinical treatment. This will be evaluated by two blinded independent reviewers through the review of pre-treatment vs. post-treatment photos taken with a VECTRA H2 (Canfield Scientific, Inc) camera.
Aggregated measurements of subcutaneous fat treatment by Cryolipolysis [Efficacy] | 12 weeks
  The primary endpoint of the study is to evaluate the efficacy of subcutaneous fat reduction in the medial intragluteal folds using the ZELTIQ System as a non-invasive clinical treatment. Quantitative measurements of efficacy will be determined by review of 3-D images from a Vectra H2 software by Canfield Scientific, Inc. measuring buttock volume difference in cc, angle formed at the inner gluteal vertex in degrees, and Height difference from the top to the bottom of the buttock in mm and surface area reduction calculations in cm2

SECONDARY OUTCOMES:
Subject satisfaction of subcutaneous fat treatment documented in written questionnaire | 12 weeks
  Subject satisfaction data will be collected at the 12-week final follow-up visit via a written questionnaire. A validated questionnaire using a likert rating scale will be utilized . Score values are 1 to 5, with high numbers meaning better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Leyda R Bowes, MD, Principal Investigator — Riverchase Dermatology
Locations (1):
- Riverchase Dermatology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be summarized based on the nature of the data. Dichotomous (e.g., gender, independent photographic review) and ordinal (e.g., Fitzpatrick Skin type) data will be tabulated by category. The mean, standard error, maximum and minimum will be tabulated for continuous data (e.g., age). The significance level will be two-sided 0.05 for all statistical tests.
Supporting Information: Study Protocol, SAP
Time Frame: May 2021 for one year
Access Criteria: Direct request to team contact listed in Ct.gov